CLINICAL TRIAL: NCT05271760
Title: Fast Track Painless Labor: New Approaches for Pain-free Delivery in Multiparous Women
Brief Title: Spinal Analgesia as Fast Track Painless Labor
Status: Completed | Type: Observational
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ahmed Abodonya, Assistant Professor, Prince Sattam Bin Abdulaziz University
Other Study IDs: REC-HSD-64-2021
Record Dates: First submitted 2021-12-08; First posted 2022-03-09 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Labor Pain; Pain, Postoperative; Pain, Acute
MeSH Terms: conditions — Labor Pain; Pain, Postoperative; Acute Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- S group: Single-shot Spinal group
  Interventions: Procedure: Single-shot spinal analgesia
- E group: Continuous Epidural
  Interventions: Procedure: Continuous epidural analgesia
- C group: combined spinal-epidural
  Interventions: Procedure: Combined spinal-epidural analgesia

INTERVENTIONS:
Procedure: Single-shot spinal analgesia — The intrathecal medication included 1ml of 0.5% heavy bupivacaine (5 mg) and 25 μg fentanyl, CSF barbotage will do to reach a total volume of 2 ml
  Groups: S group
Procedure: Continuous epidural analgesia — Epidural analgesia is performed using a 16-gauge Tuohy epidural needle using a loss-of-resistance- to-saline technique, upon feeling the loss of resistance an epidural catheter will be introduced cranially through the needle for 5 cm in the L3-L4 epidural space, after negative aspiration for blood or spinal fluid a test dose of 3 ml lidocaine 1.5% with epinephrine 1:200000 will be given via inserted catheter, 10 ml of 0.125 % bupivacaine and 2ug/ml fentanyl will be injected as a loading dose then the solution will infuse in a rate of 6 -14 ml/h.
  Groups: E group
Procedure: Combined spinal-epidural analgesia — Epidural analgesia is performed using a combined spinal-epidural set. using a loss-of-resistance- to-saline technique, upon feeling the loss of resistance, once epidural space will be detected, 27 G Whitacre spinal needle inserted through Touhy epidural needle, intrathecal injection of 1ml of 0.5% heavy bupivacaine (5 mg) and 25 μg fentanyl, CSF barbotage will do to reach a total volume of 2 ml. Then an epidural catheter will be introduced cranially through the needle for 5 cm in the L3-L4 epidural space, after negative aspiration for blood or spinal fluid.
  10 ml of 0.125 % bupivacaine and 2ug/ml fentanyl will be injected as a loading dose then the solution will infuse at a rate of 6 -14 ml/h if needed.
  Groups: C group

SUMMARY:
The purpose of this prospective, randomized, and controlled trial was to compare the efficacy of single-shot spinal analgesia to typical conventional treatments (continuous epidural analgesia and spinal-epidural combination) in reducing labor pain, particularly in multiparous women.

we will enroll in each of the three groups(S group= single-shot Spinal group), (E group= Continuous Epidural), and (C group = combined spinal-epidural) women in advanced active labor and fulfill inclusion criteria.

DETAILED DESCRIPTION:
Patients in active labor with cervical dilation between 4-5 cm multiparous with normal fetal heart rate (FHR) tracings were considered. After the request for analgesia, each patient was randomized, using a computer-generated randomization table, to receive spinal analgesia, continuous epidural analgesia, or combined spinal-epidural analgesia. Under A complete aseptic condition in a sitting position, all techniques are performed in the Labor and delivery room. All parturients are categorized into three groups as follows:

Group S (spinal n=40) The intrathecal medication included 1ml of 0.5% heavy bupivacaine (5 mg) and 25 μg fentanyl, CSF barbotage will do to reach a total volume of 2 ml. Group E (continuous Epidural n=40): Epidural analgesia is performed using a 16-gauge Tuohy epidural needle using a loss-of-resistance- to-saline technique, upon feeling the loss of resistance an epidural catheter will be introduced cranially through the needle for 5 cm in the L3-L4 epidural space, after negative aspiration for blood or spinal fluid a test dose of 3 ml lidocaine 1.5% with epinephrine 1:200000 will be given via inserted catheter, 10 ml of 0.125 % bupivacaine and 2ug/ml fentanyl will be injected as a loading dose then the solution will infuse in a rate of 6 -14 ml/h.

Group C (Combined spinal-epidural n=40) Epidural analgesia is performed using a combined spinal-epidural set. using a loss-of-resistance- to-saline technique, upon feeling the loss of resistance, once epidural space will be detected, 27 G Whitacre spinal needle inserted through Touhy epidural needle, intrathecal injection of 1ml of 0.5% heavy bupivacaine (5 mg) and 25 μg fentanyl, CSF barbotage will do to reach a total volume of 2 ml. Then an epidural catheter will be introduced cranially through the needle for 5 cm in the L3-L4 epidural space, after negative aspiration for blood or spinal fluid.

10 ml of 0.125 % bupivacaine and 2ug/ml fentanyl will be injected as a loading dose then the solution will infuse at a rate of 6 -14 ml/h if needed.

Then, the parturients will be placed in the supine position with left lateral displacement produced by placing a wedge under the right hip to prevent aortocaval compression and hypotension. Supplemental oxygen will be applied using a nasal cannula (2-4 L/min).

Each patient will receive at least 10 mL/kg Ringer lactate solution. All patients will be monitored before the procedures and every 5 minutes after for 30 for any hemodynamic instability and fetal viability The duration of analgesia is defined as the time from the injection of the local anesthetic solution until the patient requested an additional analgesic dose.

After the administration of the anesthetic solution, each patient will be evaluated by an investigator every 5 min for the first 15 min. Patients are assessed every 15 min until additional analgesia is requested.

Patient appraisal included Assessment of vital signs (blood pressure, heart rate, respiratory rate) and completion by the patient of a 10-cm linear visual analog scale (VAS) for pain (0= no pain; 10 = severe pain). Patients will be excluded from the final data analysis if the patients reported pain VAS >8 up to 15 min after the injection of the anesthetic solution. At the same time intervals, somnolence will be evaluated using a four-point ordinal scale in which 0= wide awake, 1= drowsy, 2= arousable, 3 = non-arousable, the Motor blockade will be assessed using the four-point Bromage scale. The upper level of loss of sensation to ice will be assessed in the mid-clavicular line 15 min after the injection of the anesthetic solution. Time 2 segment regressions will be assessed. Side effects such as Pruritus, nausea, or vomiting Patient and obstetrician satisfaction. All patients have continuous electronic FHR monitoring throughout labor. Any FHR abnormalities, identified by the obstetric team, will be documented. After labor, the baby will be assessed, and the mother will be nursed in a post-anesthetic care unit (PACU ) and observed if there is nausea, vomiting, dyspnea, hemodynamic changes (hypotension and reflex tachycardia), and Spo2 changes will be recorded too, also patient will be evaluated for any Sensory or motor complication. The purpose of this study is to investigate the safety and effectiveness of single-dose spinal or epidural analgesia to control labor pain in properly-selected multiparous women in a tertiary referral maternity hospital.

ELIGIBILITY:
Inclusion Criteria:

* Multiparous parturients
* ASA physical status II,
* Full-term singleton fetus
* Vertex presentation requesting analgesia during labor.
* Active labor, 4 to 5 cm dilated cervix

Exclusion Criteria:

* Patients with contraindications to regional anesthesia
* Complicated pregnancies
* Primiparous parturients
* Diagnosed fetal abnormalities
* Allergy to the study medications
* INR >1.3, and or platelets count <100,000

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: The required sample size was n= 27 in each group (Totally of 81). Therefore, we will enroll 102 patients to account for the dropout rate of 20%.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Assessment of degree of labor pain after administration of analgesia (spinal, epidural and combined spinal-epidural | 6 months
  By using Visual Analogue score (VAS score)

SECONDARY OUTCOMES:
Patient satisfaction | 6 months
  By patient satisfaction survey
Complications of technique | 6 months
  Incidence or frequency of any complication that may occur
Cost benefits | 6 months
  Cost of techniques(how much the cost of spinal kits in relation to the cost of epidural and combined spinal epidural kits in Saudi Riyal

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abodonya, MD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No